CLINICAL TRIAL: NCT01580072
Title: REgions of Europe WorkiNg toGether for HEALTH (Renewing Health)
Brief Title: Telemonitoring of Patients With COPD in Carinthia
Acronym: RenewingHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landeskrankenanstalten-Betriebsgesellschaft (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C250487
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Results first posted 2015-07-01 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive (COPD)
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

ARMS (3):
- Control group (No Intervention): Participants in the control group receive usual care.
- Self monitoring for patients with COPD (Experimental)
  Interventions: Other: self-monitoring for patients with severe COPD
- Nurse monitoring for patients with COPD (Experimental)
  Interventions: Other: nurse-monitoring for patients with severe COPD

INTERVENTIONS:
Other: self-monitoring for patients with severe COPD — Intervention Group entering vital parameters via Web Portal or automatic call center.
  Arms: Self monitoring for patients with COPD
Other: nurse-monitoring for patients with severe COPD — Nurses are entering vital parameters of the patient with mobile devices.
  Arms: Nurse monitoring for patients with COPD

SUMMARY:
Evaluation whether the introduction of large-scale telemonitoring of patients with COPD produces benefits in terms of reduced hospital readmissions, improved health related quality of life and health status. In addition, the trials evaluate the economical and organizational impact of the new services and examine their acceptability by patients and health professionals.

ELIGIBILITY:
Inclusion Criteria:

* COPD 3 or 4
* Be able to use the system provided
* Life expectancy > 12 months

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-02; Primary Completion 2013-07 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - LKH Laas, Kötschach, Carintha
  - Klinikum Klagenfurt, Klagenfurt, Carinthia
  - LKH Villach, Villach, Carinthia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to organisational changes in the participating home nursing organisation and due to the age of the patients no nurse monitoring patients were admitted. Furthermore a first examination in the hospitals seemed to be hindering for these patients.
Period: Overall Study
Arm/Group | Control Group | Self Monitoring for Patients With COPD | Nurse Monitoring for Patients With COPD
Started | 28 | 37 | 0
Completed | 16 | 28 | 0
Not Completed | 12 | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Self Monitoring for Patients With COPD | Nurse Monitoring for Patients With COPD | Total
Number analyzed (Participants) | 28 | 37 | 0 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.62 (10.28) | 63.83 (7.69) |  | 68.04 (8.80)
Gender [Number; unit: participants]
  Female | 10 | 11 |  | 21
  Male | 18 | 26 |  | 44
Region of Enrollment [Number; unit: participants]
  Austria | 28 | 37 |  | 65

OUTCOME MEASURES:

1. Primary Outcome: Health Related Quality of Life as Measured by the Short-Form 36 Version 2 Questionnaire; The Short Form (36) Health Survey is a 36-item, Patient-reported Survey of Patient Health. The SF-36 is a Measure of Health Status.
Description: Baseline analyses and analyses after 12 months were conducted. Normal distribution is not given for SF-36 scales, means and Standard Deviation are reported. A high score defines a more favorable health state, items are scored on a 0 to 100 range. Scale scores represent the average for all items in the scale that the respondent answered.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Self Monitoring for Patients With COPD | Nurse Monitoring for Patients With COPD
Number analyzed (Participants) | 16 | 28 | 0
units on a scale
  physical functioning baseline | 35.0 (27.4) | 48.2 (24.5) |
  physical functioning after 12 months | 22.8 (15.4) | 39.8 (31.5) |
  role physical baseline | 19.5 (19.2) | 40.7 (20.0) |
  role physical after 12 months | 28.9 (20.9) | 35.9 (25.0) |
  bodily pain baseline | 59.1 (40.2) | 55.6 (28.8) |
  bodily pain after 12 months | 52.8 (39.1) | 55.3 (32.6) |
  general health baseline | 40.1 (26.7) | 49.3 (14.4) |
  general health after 12 months | 36.3 (21.3) | 47.3 (25.1) |
  vitality baseline | 38.3 (25.1) | 44.0 (16.4) |
  vitality after 12 months | 35.5 (22.4) | 44.6 (27.9) |
  social functioning baseline | 58.6 (36.7) | 67.4 (24.4) |
  social functioning after 12 months | 64.1 (36.8) | 61.2 (33.9) |
  role emotional baseline | 27.6 (28.7) | 53.4 (28.8) |
  role emotional after 12 months | 45.8 (29.0) | 53.7 (33.6) |
  mental health baseline | 53.1 (26.6) | 59.5 (19.9) |
  mental health after 12 months | 56.6 (27.8) | 59.6 (26.7) |
  physical component score baseline | 35.3 (11.3) | 38.1 (7.6) |
  physical component score after 12 months | 31.0 (9.2) | 36.1 (10.3) |
  mental component score baseline | 35.0 (13.1) | 41.8 (11.7) |
  mental component score after 12 months | 41.0 (14.6) | 42.7 (14.8) |

2. Primary Outcome: Number of Inpatient Stays
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: inpatient stays
Arm/Group | Control Group | Self Monitoring for Patients With COPD | Nurse Monitoring for Patients With COPD
Number analyzed (Participants) | 28 | 37 | 0
inpatient stays | 1.54 (2.27) | 1.16 (1.91) |

3. Secondary Outcome: Number of Bed Days for Hospitalised Patients
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: bed days
Arm/Group | Control Group | Self Monitoring for Patients With COPD | Nurse Monitoring for Patients With COPD
Number analyzed (Participants) | 28 | 37 | 0
bed days | 6.87 (6.78) | 4.92 (6.36) |

4. Secondary Outcome: Number of Primary Care Visits
Description: Not all data were available, so only participants with consistent data were taken into comparison, this lead to a lower number of patients in this outcome measurement.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: visits GP
Arm/Group | Control Group | Self Monitoring for Patients With COPD | Nurse Monitoring for Patients With COPD
Number analyzed (Participants) | 19 | 30 | 0
visits GP | 13.21 (10.27) | 9.67 (10.09) |

5. Secondary Outcome: Number of Specialist Visits
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: visits specialists
Arm/Group | Control Group | Self Monitoring for Patients With COPD | Nurse Monitoring for Patients With COPD
Number analyzed (Participants) | 19 | 30 | 0
visits specialists | 3.31 (3.15) | 4.6 (5.03) |

6. Secondary Outcome: Number of Consultations of Emergency Doctor
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: consultations ED
Arm/Group | Control Group | Self Monitoring for Patients With COPD | Nurse Monitoring for Patients With COPD
Number analyzed (Participants) | 19 | 30 | 0
consultations ED | 0.79 (1.03) | 1.17 (2.42) |

7. Secondary Outcome: All Cause Mortality
Description: deceased patients in respect to participating patients, by obituary column
Time Frame: 12 months
Reporting Status: Not Posted

8. Secondary Outcome: COPD Assessment Test CAT (Carinthia)
Description: No data available
Time Frame: 12 months
Reporting Status: Not Posted

9. Secondary Outcome: St. George's Respiratory Questionnaire SGRQ (Carinthia)
Description: The SGRQ is a 50-item questionnaire developed to measure health status (quality of life) in patients with diseases of airways obstruction.
  Scores are calculated for three domains:
  Symptoms, Activity and Impacts as well as a total score. Psychometric testing has demonstrated its repeatability, reliability and validity. Sensitivity has been demonstrated in clinical trials.
  A minimum change in score of 4 units was established as clinically relevant after patient and clinician testing. The SGRQ has been used in a range of disease groups including asthma, chronic obstructive pulmonary disease (COPD) and bronchiectasis, and in a range of settings such as randomised controlled therapy trials and population surveys.Due to missing data not all questoinnaires could be taken into consideration. Normal distribution is not given for SGRQ scales; Scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best pos
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Self Monitoring for Patients With COPD | Nurse Monitoring for Patients With COPD
Number analyzed (Participants) | 16 | 25 | 0
units on a scale
  sympoms score baseline | 74.0 (20.1) | 69.0 (18.0) |
  sympoms score after 12 months | 67.4 (24.2) | 61.2 (27.6) |
  activity score baseline | 76.3 (17.2) | 68.9 (22.9) |
  activity score after 12 months | 79.3 (13.5) | 62.4 (28.4) |
  impacts score baseline | 55.1 (17.9) | 42.6 (20.9) |
  impacts score after 12 months | 54.3 (20.1) | 42.3 (23.3) |
  total score baseline | 64.8 (15.3) | 54.6 (18.1) |
  total score after 12 months | 64.2 (17.7) | 50.8 (24.0) |

10. Secondary Outcome: BODE Index (Carinthia)
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control Group | Self Monitoring for Patients With COPD | Nurse Monitoring for Patients With COPD
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/37 | 0/0
Other Adverse Events (participants affected / at risk) | 0/28 | 0/37 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes